CLINICAL TRIAL: NCT05351073
Title: The Safety and Feasibility of Normobaric Oxygen Administration for SUSPEcted Acute Stroke uNder Pre-hoSpItal cONdition--A Pilot Trial
Brief Title: The Prehospital Administration of Normobaric Oxygen in Suspected Stroke
Acronym: NO SUSPENSION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO-SUSPENSION
Record Dates: First submitted 2022-02-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Acute Stroke; Ischemic Stroke, Acute
Keywords: Acute stroke; Normobaric oxygen; Stroke neuroprotection
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normobaric Oxygen Inhalation Group (Experimental): Participants in the intervention group will receive oxygen inhalation through a mask at a rate of 10 L/min at 1 absolute atmosphere pressure (1 ATA = 101.325 kPa) after randomization until adimisson to the hospital. Participants will subsequently receive standard diagnosis and treatment service according to the guidelines during hospitalization.
  Interventions: Drug: NBO
- Control Group (No Intervention): Participants in the control group will not receive oxygen inhalation therapy during ambulance transportation. Participants will subsequently receive standard diagnosis and treatment service according to the guidelines during hospitalization.

INTERVENTIONS:
Drug: NBO — Oxygen inhalation through a mask at a rate of 10 L/min at 1 absolute atmosphere pressure (1 ATA = 101.325 kPa)
  Arms: Normobaric Oxygen Inhalation Group

SUMMARY:
The primary purpose of this study is to explore the feasibility and safety of normobaric oxygen therapy (NBO) under pre-hospital condition in patients with suspected stroke.

DETAILED DESCRIPTION:
Despite the application of thrombolytic drugs and endovascular treatment, there is still a gap between the successful recanalization and ideal clinical outcomes for stroke patients. Neuroprotective treatment is considered as a promising adjuvant to ameliorate this situation. Previous researches demonstrated the neuroprotective effects of Normobaric Hyperoxia (NBO) in animal models from multiple perspectives. Moreover, NBO is distinctive for its ubiquity, conveniency, high compatibility, and wide adaptability, making it superior to other neuroprotective interventions in a pre-hospital setting. Therefore, the investigators conducted this pilot study to further explore the feasibility and safety of NBO under a pre-hospital condition in patients with suspected stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. Suspected stroke screened by the "Gaze- Face Arm Speech Time" scale (G-FAST score ≥ 1).
3. Within 24 hours of symptom onset
4. SpO2 > 94%.

Exclusion Criteria:

1. Coma: Glasgow coma score (GCS) < 8.
2. Hypoglycemia: Blood glucose < 2.8mmol /L.
3. Known history of seizure.
4. Recent stroke or brain trauma within past 30 days.
5. Previous Modified Rankin Scale (mRS) ≥2.
6. Rapid improvement of neurological dysfunction (deficit present less than 15 min).
7. Unstable vital signs.
8. Known respiratory distress, respiratory dysfunction, or any contraindications to high-flow oxygen inhalation therapy.
9. Patient unable to cooperate with the trial procedure.
10. Any condition which might increase the risk to the patient in the judgment of the investigator.
11. Patient or available legally authorized representative unable to provide written or witnessed oral consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Time intervals of the prehospital transportation process | Day 1
  Time intervals between stroke onset, paramedic arrival on the scene, the departure from the scene, and admission to the hospital emergency department.

SECONDARY OUTCOMES:
Safety Outcome | Day 1
  Incidence of adverse events during oxygen inhalation reported by the ambulance nurses.
Recruitment rate | From the date of recruitment initiation until the date of recruitment completion, assessed up to 24 months.
  The rate of patients successfully recruited to the trial by prehospital paramedics.
Final diagnosis | From the date of recruitment initiation until the date of recruitment completion, assessed up to 24 months.
  The final diagnosis of the patients enrolled in the trial.
Plateletto-lymphocyte ratio(PLR) | Day1
  The platelet-to-lymphocyte ratio (PLR) is calculated as the absolute count of platelet divided by the absolute count of lymphocytes.
Systemic immune-inflammation index (SII) | Day 1
  Systemic immune-inflammation index (SII) is calculated with the formula SII = (Peripheral platelet counts× Neutrophil counts)/Lymphocyte counts.
Neutrophil-to-lymphocyte ratio (NLR) | Day 1
  Neutrophil to lymphocyte ratio (NLR) is calculated as the absolute count of neutrophils divided by the absolute count of lymphocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes